CLINICAL TRIAL: NCT01076478
Title: Asian Study on Cilostazol Effectivity in Neuropathies of Diabetes Mellitus Type 2-A Pilot Study in the Philippines
Acronym: ASCEND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical, Inc., Philippines (Industry)
Responsible Party: Evelio Valdes/CRA, Otsuka Pharmaceutical, Inc., Philippines
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLT-004-01
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Polyneuropathy
Keywords: Symmetric Diabetic Polyneuropathy
MeSH Terms: conditions — Polyneuropathies | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Placebo Comparator): 2 tablets BID
  Interventions: Drug: Cilostazol
- Arm 2 (Experimental): 100 mg Cilostazol (2 tablets BID)
  Interventions: Drug: Cilostazol
- Arm 3 (Experimental): 200 mg Cilostazol (2 Tablets BID)
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Cilostazol — 100 mg, 200mg tablet Cilostazol
  Other Names: Cilostazol, Pletaal, Pletal

SUMMARY:
To describe if there are differences in the subjective, objective and electrophysiologic parameters of diabetic polyneuropathies at baseline, four (4) weeks, eight (8) weeks, and twelve (12) weeks after Cilostazol therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent 2. Male and Female ages 18 to 70 years old. To be able to eliminate Type I Diabetes Mellitus among the younger subjects, we will only recruit patients who are stable on oral hypoglycemic agent. 3. Established diagnosis of diabetes mellitus type 2 (National Diabetes Data Group) who are currently on good control of the diabetic state.

4. Presence of predominantly distal symmetrical sensory polyneuropathy of the lower limbs as assessed by NSS, NIS and NCS.

Exclusion Criteria:

1. Current use of potentially neuropathic agents (Isoniazid, Phenytoin, Dapsone, Metronidazole, Vinca Alkaloids, etc.) within the past 1 month;
2. Presence of severe metabolic disease (renal failure, hepatic failure, etc.), alcoholism and malignancy;
3. Presence of hemorrhagic tendencies;
4. Patients who are diagnosed to be of Type 1 Diabetes Mellitus;
5. Pregnant and lactating patients, including those who plan to have pregnancy within the study period.
6. Concomitant intake of agents currently used to treat neuropathic pain like gabapentin, carbamazepine/ oxcarbazepine, anti-depressants (tricyclic anti-depressants and SSRIs) and topical capsaicin.
7. Concomitant intake of other anti-platelet agents, rheologic agents and anticoagulants.
8. Have received Cilostazol therapy within the past three (3) months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-03; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Subjective neuropathy assessment by NSS (Neuropathy Symptom Scores)from Baseline (BS) to week 12 (W12) after Cilostazol therapy of the three (3) arms of the study. | 12 weeks
Objective neuropathy assessment by NIS (Neuropathy Impairment Scores)from Baseline (BS) to week 12 (W12) after Cilostazol therapy of the three (3) arms of the study. | 12 weeks
Electrophysiologic assessment by NCS (Nerve Conduction Studies) from Baseline (BS) to week 12 (W12) after Cilostazol therapy of the three (3) arms of the study. | 12 weeks
To determine the relationship of peripheral neuropathy with peripheral vascular disease using the WIQ and the ABI from baseline to W12. | 12 weeks

SECONDARY OUTCOMES:
To determine if there is improvement in subjective parameters of neuropathy as assessed by NSS and NSC (Neuropathy Symptoms and Change Questionnaire) from baseline to week 4 (W4), week 8 (W8) and week 12 (W12) after Cilostazol therapy. | 12 weeks
To determine if there is improvement in objective parameters using NIS and NCS from baseline to W4, W8 and W12 after Cilostazol therapy. | 12 weeks
To compare the effectivity of low dose (100mg) and high dose (200mg) Cilostazol based on subjective (NSS, NSC) and objective parameters (NIS, NCS) from baseline, to W4, W8 and W12. | 12 weeks
To assess the safety of Cilostazol therapy. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Rosales, MD, PhD, Principal Investigator — University of Santo Tomas Hospital
Locations (1):
- University of Santo Tomas Hospital, Manila, Philippines